CLINICAL TRIAL: NCT03681158
Title: An Open-label Study of Excretion Balance and Pharmacokinetics Following a Single Oral Dose of [14C]-Sodium Valproate (3.7 MBq) in Healthy Postmenopausal or Permanently Sterile Female Subjects
Brief Title: Study of Excretion Balance and Pharmacokinetics of [14C]-Sodium Valproate (3.7 MBq) in Healthy Postmenopausal or Permanently Sterile Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEX15316; 2017-004987-36 (EudraCT Number); U1111-1205-1651 (Other: UTN)
Record Dates: First submitted 2018-09-14; First posted 2018-09-21 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sodium valproate (Experimental): Single oral dose of sodium valproate containing [14C]-sodium VPA
  Interventions: Drug: sodium valproate

INTERVENTIONS:
Drug: sodium valproate — Pharmaceutical form:Powder for oral solution reconstituted with water Route of administration: Oral
  Other Names: LA40220

SUMMARY:
Primary Objectives:

* To determine the excretion balance and systemic exposure of radioactivity after oral administration of [14C]-sodium valproate (VPA) .
* To determine the pharmacokinetics of sodium VPA and metabolite(s) and its contribution to the overall exposure of radioactivity.
* To collect samples in order to determine the metabolic pathways of sodium VPA and identify the chemical structures and main excretion route of the main metabolites.

Secondary Objective:

To assess the clinical and biological tolerability of oral solution of sodium VPA.

DETAILED DESCRIPTION:
Total study duration is 3 to 10 weeks, including a screening period of 8 to 28 days, treatment period of up to 15 days and a follow-up and end of study of up to 4 weeks.

ELIGIBILITY:
Inclusion criteria :

* Female subjects, between 30 and 60 years of age, inclusive.
* Body weight between 40.0 and 90.0 kg, inclusive, body mass index between 18.0 and 30.0 kg/m2, inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal vital signs after 10 minutes resting in supine position: 95 mmHg < systolic blood pressure (SBP) <140 mmHg or, for subjects over 45 years of age, <150 mmHg, 45 mmHg < diastolic blood pressure (DBP) <90 mmHg, 40 bpm < heart rate (HR) <100 bpm
* Standard 12-lead electrocardiogram (ECG) parameters after 10 minutes resting in supine position in the following ranges; 120 ms<PR<220 ms, QRS<120 ms, QTc≤450 ms and normal ECG tracing unless the Investigator considers an ECG tracing abnormality to be not clinically relevant, or for subjects over 45 years of age, standard 12-lead ECG without clinically significant abnormality, in the judgment of the Investigator, with QTc≤470 ms.
* Laboratory parameters within the normal range (or defined screening threshold for the Investigator site), unless the Investigator considers an abnormality to be clinically irrelevant for healthy subjects; however, serum creatinine, alkaline phosphatase, hepatic enzymes (aspartate aminotransferase, alanine aminotransferase), and total bilirubin (unless the subject has documented Gilbert syndrome) should not exceed the upper laboratory norm.
* Surgically and permanently sterile (hysterectomy, bilateral salpingectomy or bilateral salpingo-oophorectomy) at least 3 months earlier or postmenopausal. Menopause is defined as being amenorrheic for at least 2 years with plasma FSH level > 30 UI/L. No additional contraception is required.
* Having given written informed consent prior to undertaking any study-related procedure.
* Covered by a health insurance system where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research.
* Not under any administrative or legal supervision.
* Normal renal function as expressed by a creatinine clearance > 80 mL/min as calculated by the Cockroft and Gault formula

Exclusion criteria:

* Any subject with specific dietary habits, such as vegan.
* Any subject with irregular bowel habits (more than 3 bowel movements/day or less than 1 every 2 days).
* Any subject undergoing dental care or presenting with dental caries.
* Any subject who is occupationally exposed to radiation as defined in the Ionising Radiations Regulations 2017.
* Participation in a trial with 14C-radiolabelled medication in the 12 months preceding the study.
* Radiation exposure, including that from the present study and radiopharmaceuticals or radionuclides in therapeutic or diagnostic procedures, but excluding background radiation, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years.
* Poor metabolizer status for CYP2C9, CYP2C19, CYP2D6 (by genotyping).
* Any consumption of citrus (grapefruit, orange, etc) or their juices within 5 days before inclusion.
* Any contra-indications to sodium VPA according to the applicable labeling (including personal or family history of severe hepatic dysfunction, urea cycle disorders, porphyria, hypersensitivity to valproate, active liver disease, pregnancy, child bearing potential) and patients known to have mitochondrial disorders caused by mutations in the nuclear gene encoding mitochondrial enzyme polymerase γ (POLG, e.g. Alpers-Huttenlocher Syndrome).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Percentage of radioactive dose excreted in urine and feces | Day 1 to Day 43
  Fractional and cumulative percentage of radioactive dose excreted in urine and feces
Assessment of key metabolite(s) of sodium valproate | Day 1 to Day 43
  key metabolite(s) of sodium valproate will be assessed in plasma, urine and feces.
Assessment of PK parameters: Cmax | Day 1 to 8, Day 12 to Day 15, Day 22, Day 29, Day 36, Day 43
  Maximum plasma or blood concentration observed
Assessment of PK parameters: tmax | Day 1 to 8, Day 12 to Day 15, Day 22, Day 29, Day 36, Day 43
  Time to reach Cmax (tmax)
Assessment of PK parameters: AUClast | Day 1 to 8, Day 12 to Day 15, Day 22, Day 29, Day 36, Day 43
  Area under the plasma concentration versus time curve calculated from time zero to the real time, tlast (time corresponding to the last concentration above the limit of quantification, Clast (AUClast)
Assessment of PK parameters: AUC | Day 1 to 8, Day 12 to Day 15, Day 22, Day 29, Day 36, Day 43
  Area under the plasma concentration versus time curve extrapolated to infinity (AUC)
Assessment of PK parameters: t1/2z | Day 1 to 8, Day 12 to Day 15, Day 22, Day 29, Day 36, Day 43
  Terminal half-life associated with the terminal slope (λz) (t1/2z) in plasma, blood radioactivity and plasma VPA
Assessment of PK parameters: B/P (blood/plasma radioactivity ratio) | Day 1 to 8, Day 12 to Day 15, Day 22, Day 29, Day 36, Day 43
  Blood to plasma radioactivity ratio calculated at each time point
Assessment of PK parameters: RCmax (VPA to radioactivity ratio for plasma Cmax) | Day 1 to 8, Day 12 to Day 15, Day 22, Day 29, Day 36, Day 43
  RCmax is calculated as Cmax(VPA)/Cmax (radioactivity)
Assessment of PK parameters: RAUC (VPA to radioactivity ratio for plasma AUC) | Day 1 to 8, Day 12 to Day 15, Day 22, Day 29, Day 36, Day 43
  RAUC is calculated as AUC(VPA)/AUC (radioactivity)

SECONDARY OUTCOMES:
Safety- Adverse Events | From day -1 to 43
  Adverse events, spontaneously reported by the subject or observed by the Investigator from day -1 to day 43

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site number, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org